CLINICAL TRIAL: NCT03432923
Title: A Multi-center, Double-blind, Randomized, Parallel-group, Placebo-controlled Study to Determine the Efficacy and Safety of a Benzocaine Lozenge for Treatment of Sore Throat Caused by URTI in Adults.
Brief Title: A Study to Determine the Efficacy and Safety of a Benzocaine Lozenge for Treatment of Sore Throat.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McNeil AB (Industry)
Collaborators: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CO-161004120104-URCT; 129649CGH3001 (Other: Janssen Pharmaceutica NV)
Record Dates: First submitted 2018-01-23; First posted 2018-02-14 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Sore Throat
MeSH Terms: conditions — Pharyngitis | interventions — Benzocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind design. Placebo indistinguishable to active in appearance and dosing schedule.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Benzocaine 8 mg (Experimental): Benzocaine 8 mg, oval, white to slightly beige to yellow film coated tablet. One lozenge to be dissolved slowly in the mouth every 2 hours. Max 6 per day, max treatment 5 days.
  Interventions: Drug: Benzocaine 8 mg
- Placebo (Placebo Comparator): Placebo, oval, white to slightly beige to yellow film coated tablet. One lozenge to be dissolved slowly in the mouth every 2 hours. Max 6 per day, max treatment 5 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Benzocaine 8 mg — Benzocaine 8 mg, oval, white to slightly beige to yellow film coated tablet. One lozenge to be dissolved slowly in the mouth every 2 hours. Max 6 per day, max treatment 5 days.
  Other Names: Benzocaine lozenge
  Arms: Benzocaine 8 mg
Drug: Placebo — Placebo, oval, white to slightly beige to yellow film coated tablet. One lozenge to be dissolved slowly in the mouth every 2 hours. Max 6 per day, max treatment 5 days.
  Other Names: Placebo lozenge
  Arms: Placebo

SUMMARY:
A multi-center, double-blind, randomized, parallel-group, placebo-controlled study to determine the efficacy and safety of a benzocaine lozenge for symptomatic treatment of sore throat caused by acute upper respiratory tract infection in adults.

DETAILED DESCRIPTION:
This multi-center, double-blind, randomized, parallel-group, placebo-controlled study consists of two parts, an initial efficacy and safety part performed at the clinic on the first treatment day and a safety follow up home-use treatment part with an intermediate site visit.

Following screening and randomization, subjects suffering from throat pain caused by an acute upper respiratory tract infection will receive a single dose of study medication, benzocaine 8 mg or placebo lozenge, and will be followed for a 3 hour assessment period where primary and secondary efficacy measurements will be collected.

Onset and duration of what the subject consider to be perceptible and meaningful pain relief, respectively, will be measured by collecting time point for reported onset in relation to time of intake of the single dose.

The subjects will assess their pain intensity and the degree of difficulty swallowing during multiple assessment time points throughout the 3 hour period on 11-point numerical rating scales (NRS) where 0=no pain/not difficult, 10=very severe pain/very difficult.

The subjects will rate their sore throat condition in a subject questionnaire at baseline and after 2 and approximately 72 hours of treatment. The subjects will also rate how satisfied they were with the assigned study medication as a treatment for sore throat in a global evaluation assessment at the end of the 3 hour assessment period and after approximately 72 hours of treatment.

After initiation of treatment and the initial efficacy part of the study (Day 1), the subjects will be released for home based treatment according to label to complete the safety part of the study. The subjects will be equipped with study medication according to randomization and diaries to record number of study medication doses taken per day. The subjects will be instructed to follow their respective treatment label and return to the site for safety follow up at study Day 4 (target approximately 72 hours of treatment) and at the end of treatment, at Day 6 (target approximately 120 hours of treatment).

ELIGIBILITY:
Subject Inclusion Criteria

Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study:

1. Subjects of 18 years of age or older, suffering from throat pain caused by acute upper respiratory tract infection;
2. Symptoms of acute throat pain have been persisting for minimum of 3 hour and maximum 72 hours;
3. Have body mass index (BMI) 18.5 to 35 (inclusive) at screening;
4. Indicate at least a score of 5 on an 11-point (0-10) pain intensity numerical rating scale (PI-NRS) at screening and at baseline;
5. Females of childbearing potential must have a negative urine pregnancy test at screening;
6. Male and non-pregnant, non-lactating female agree to the contraceptive requirements (including female partner´s use of highly effective form of birth control for at least 3 months before the study, during the study and up to 30 days after the last dose of investigational product) as outlined in protocol.
7. Are able and willing to comprehend and follow the requirements of the study (including availability on scheduled visit dates) based upon research site personnel´s assessment;
8. Are able to read and understand the local language;
9. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study and consents to participate.

Subject Exclusion Criteria

Subjects presenting with any of the following will not be included in the study:

1. Are female and who are pregnant, breastfeeding or intended pregnancy;
2. Are male with a pregnant partner or a partner who is currently trying to become pregnant;
3. Have a known allergy or hypersensitivity to benzocaine or any of the excipients of the formulations;
4. Known or suspected NADH-diaphorase deficiency;
5. Presence or history of medical condition in the investigator's opinion that may jeopardize the subject's safety or well-being, or the integrity of the study (e.g., hepatic, renal, pancreatic, gastrointestinal, cardiovascular, cerebrovascular, thyroid, seizure, asthma, allergy, drug intolerance, or psychiatric disorders; uncontrolled hypertension indicated as systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg; or uncontrolled diabetes in the last 6 months);
6. Suspected alcohol or substance abuse (e.g., amphetamines, benzodiazepines, cocaine, marijuana, opiates);
7. Clinically significant laboratory abnormality that cannot be explained by the acute upper respiratory tract infection. Subjects with increased glucose level after a meal are eligible if there is no uncontrolled diabetes in last 6 months, but not eligible if increased glucose level in a fasted state;
8. Presenting axillary temperature of 38.5 Celsius degrees or above;
9. Acute and/or chronic respiratory tract disease or other concomitant disease with potential to compromise breathing (asthma, bronchopneumonia, bronchitis);
10. Blood dyscrasias or suspected fungal upper respiratory tract infection e.g., candida infection;
11. Known or suspected bacterial upper respiratory tract infection or purulent pharyngitis;
12. Known or suspected diphtheria or clinical signs of active herpes infection;
13. Positive result in express throat test for Streptococcus;
14. Known or suspected pneumonia as verified with chest X-ray examination;
15. Routine use of oral analgesics, and/or NSAIDs ≥5 times per week. If routine use is stopped, a wash out period of at least 24 hours should have been passed since the last dose;
16. Treatment with steroids, oro-pharyngeal therapeutic agents, anticonvulsants, psychotropic or immunosuppressant agents within 8 hour (or with prolonged action NSAIDs within 10 days) or antibiotics within 14 days up to first dose;
17. Use on any confectionery lozenge/tablet/gum or any products with demulcent properties within previous 2 hour prior to first dose;
18. Use of any analgesic, oral anesthetics, antipyretic or "cold" medication within previous 8 hour, for Naproxen containing products within previous 12 hour prior to first dose;
19. Use of any antiseptics and/or oral rinses (e.g., Hexetidine, Listerine, Myramistin) within previous 2 hours prior to first dose;
20. Participate in any interventional clinical studies within 30 days before screening or had participated in this current study previously;
21. Subjects who are related to those persons involved directly or indirectly with the conduct of this study (i.e., principal investigator, sub-investigators, study coordinators, other site personnel, employees of Sponsor (including group of Johnson & Johnson companies) subsidiaries, contractors of Sponsor (including group of Johnson & Johnson companies), and the families of each).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2018-04-21 (Actual); Study Completion 2018-04-21 (Actual)

PRIMARY OUTCOMES:
Time to meaningful pain relief. | 3 hours
  A timer is started upon the intake of a single dose and stopped when the subject considers he/she has experienced meaningful pain relief.

SECONDARY OUTCOMES:
Time to perceptible pain relief (onset of therapeutic effect). | 3 hours
  A timer is started upon the intake of a single dose and stopped when the subject considers he/she has experienced perceptible pain relief.
Change from baseline in sore throat pain intensity self-ratings at 2.5, 5, 7.5, 10 and 15 min after intake, respectively. | 15 minutes
  Change from baseline in sore throat pain intensity self-ratings at 2.5, 5, 7.5, 10 and 15 min after intake, respectively.
Mean change from baseline in sore throat pain intensity self-ratings based on all assessments up to 15, 30, 60, 120, and 180 min after intake as well as during the second (60+ to 120 min) and third hour (120+ to 180 min) after intake, respectively. | 3 hours
  Mean change from baseline in sore throat pain intensity self-ratings based on all assessments up to 15, 30, 60, 120, and 180 min after intake as well as during the second (60+ to 120 min) and third hour (120+ to 180 min) after intake, respectively.
Change from baseline in self-ratings of difficulty swallowing at 2.5, 5, 7.5, 10 and 15 min after intake, respectively. | 15 minutes
  Change from baseline in self-ratings of difficulty swallowing at 2.5, 5, 7.5, 10 and 15 min after intake, respectively.
Mean change from baseline in self-ratings of difficulty swallowing based on all assessments up to 15, 30, 60, 120, and 180 min after intake as well as during the second (60+ to 120 min) and third hour (120+ to 180 min) after intake, respectively. | 3 hours
  Mean change from baseline in self-ratings of difficulty swallowing based on all assessments up to 15, 30, 60, 120, and 180 min after intake as well as during the second (60+ to 120 min) and third hour (120+ to 180 min) after intake, respectively.
Continuous period of time within the 3 hour test period with perceptible pain relief. | 3 hours
  Continuous period of time within the 3 hour test period with perceptible pain relief.
Continuous period of time within the 3 hour test period with meaningful pain relief. | 3 hours
  Continuous period of time within the 3 hour test period with meaningful pain relief.
Change from baseline in self-ratings, referring to the time period since start of treatment, of the extent to which the sore throat condition diverts the subject's concentration, assessed after 2 and 72 hour of treatment, respectively. | 72 hours
  Change from baseline in self-ratings, referring to the time period since start of treatment, of the extent to which the sore throat condition diverts the subject's concentration, assessed after 2 and 72 hour of treatment, respectively.
Change from baseline in self-ratings, referring to the time period since start of treatment, of the extent to which the sore throat condition makes it difficult for the subject to speak, assessed after 2 and 72 hour of treatment, respectively. | 72 hours
  Change from baseline in self-ratings, referring to the time period since start of treatment, of the extent to which the sore throat condition makes it difficult for the subject to speak, assessed after 2 and 72 hour of treatment, respectively.
Subject ratings with respect to the degree of experienced improvement in their sore throat condition, assessed after 2 and 72 hour of treatment, respectively. | 72 hours
  Subject ratings with respect to the degree of experienced improvement in their sore throat condition, assessed after 2 and 72 hour of treatment, respectively.
Subject ratings with respect to the extent to which they were able to forget their sore throat condition, assessed after 2 and 72 hour of treatment, respectively. | 72 hours
  Subject ratings with respect to the extent to which they were able to forget their sore throat condition, assessed after 2 and 72 hour of treatment, respectively.
Subject ratings with respect to the degree of overall satisfaction with their assigned study medication for sore throat, rated at the end of the 3 hour assessment period and 72 hours of treatment, respectively. | 72 hours
  Subject ratings with respect to the degree of overall satisfaction with their assigned study medication for sore throat, rated at the end of the 3 hour assessment period and 72 hours of treatment, respectively.
Frequency and severity of treatment emergent AEs reported during the study | Through study completion, an average of 5 months.
  Frequency and severity of treatment emergent AEs reported during the study
Frequency and severity of AEs possibly, probably, or very likely related to the study drug during study treatment | Through study completion, an average of 5 months
  Frequency and severity of AEs possibly, probably, or very likely related to the study drug during study treatment
Occurrence of serious AEs (SAEs), and AEs resulting in pre-mature withdrawal from the study | Through study completion, an average of 5 months.
  Occurrence of serious AEs (SAEs), and AEs resulting in pre-mature withdrawal from the study

OTHER OUTCOMES:
Subject compliance with the study medication dosing regimen by reporting of doses taken in subject diary. | Through study completion, an average of 5 months.
  Subject compliance with the study medication dosing regimen by reporting of doses taken in subject diary.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Sacavage, Study Director — Medical Affairs and Clinical Research
Locations (19):
- Russia (19):
  - Railway Clinical Hospital n.a. N.A. Semashko Lyublino railway station of the Russian Railways, Stavropolskaya str., 23, build.1,, Moscow
  - City Clinical Hospital n.a. V.M. Buyanov Bakinskaya str., 26, Moscow
  - Central Clinical Hospital of Russian Academy of Sciences Litovskiy bulvar, 1A, Moscow
  - Federal State Budgetary Institution "Policlinic #5" of Administrative Department of the President of the Russian Federation Plyushchikha str., 14, Moscow
  - Unimed-C 26 Bakinskikh Komissarov str., 11, Moscow
  - Clinic of the Modern Medicine Pobedy ploshad, 2, bldg. 1, Moscow
  - State Budgetary Healthcare Institution City Clinical Hospital n.a. M.E. Zhadkevich, Moscow
  - Hospital of Russian Academy of Sience Oktyabrskiy prospect, 3, Moscow
  - International Medical Centre SOGAZ Malaya Konushennaya str., 8A, Saint Petersburg
  - " City Polyclinic #25 of the Nevsky District of SPB" Prospekt Solidarnosti, 1, bldg 1, litera "А", Saint Petersburg
  - Clinical Hospital of Russian Academy of Sciences Morisa Toreza str., 72, Saint Petersburg
  - LLC "Medical Center "Reavita Med SPb" Uchebniy per., 2, Saint Petersburg
  - OOO Medpomoshch " Medicaid LLC" Vyborgskoe shosse, 5, bldg. 1, Saint Petersburg
  - Medical Research Institute LLC Koli Tomchaka str., 25, Saint Petersburg
  - Eco-safety Ltd Prospekt Gagarina, 65, Saint Petersburg
  - City Out-Patient Clinic #51 Prospekt Kosmonavtov, 35, Saint Petersburg
  - LLC Kurator Krasnoputilovskaya str., 125, Saint Petersburg
  - BioEq, LLC "Lit. Zh, 23, Krasnogvardejskiy per., Saint Petersburg
  - St. Petersburg SBHI City Hospital #40, 9 letter B, Borisova str, Saint Petersburg

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CO-161004120104-URCT&attachmentIdentifier=dfaaae21-b504-4e13-90a5-e47bb650c5fb&fileName=CSR_CO-161004120104-URCT-Section_2_-_Synopsis.pdf&versionIdentifier=